CLINICAL TRIAL: NCT00044148
Title: The Effect of LY333531 on Albuminuria in Patients With Type 2 Diabetes A Pilot Clinical Trial
Brief Title: The Effect of LY333531 on Protein in the Urine in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chromaderm, Inc. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 6249; B7A-MC-MBDA
Record Dates: First submitted 2002-08-20; First posted 2002-08-21 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Diabetic Nephropathy
Keywords: Persistent Albuminuria
MeSH Terms: conditions — Diabetic Nephropathies | interventions — ruboxistaurin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: LY333531

SUMMARY:
The purpose of this study are to determine 1) Whether Ly333531 can reduce urinary albumin/creatinine excretion in patients with Type II diabetes and persistent albuminuria 2) Whether LY333531 reduces urinary TGF-B, 3) the safety of LY333531 and any side effects that may be associated with it.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Greater than or equal to 30 years of age
* Albumin to Creatinine ratio (greater than 200 mg/g and less than 2000 mg/g) 4)Without language barrier.

Exclusion Criteria:

* Serum Creatinine greater than 2.0 mg/dl males or greater than 1.7 mg/dl females
* B/P greater than 150 systolic and greater than 90 diastolic
* Hemoglobin Alc greater than 11%
* Liver Function Tests 2 times upper limit of normal
* Poor medical or psychiatric risk.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2002-07-16 (Actual); Primary Completion 2004-04-28 (Actual); Study Completion 2004-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - La Jolla, California
  - Walnut Creek, California
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Waltham, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Greenville, North Carolina
  - Dallas, Texas
  - Seattle, Washington
  - Spokane, Washington